CLINICAL TRIAL: NCT05181904
Title: Gastric Content Ultrasound Monitoring Prior to Extubation in Critically Ill Children
Acronym: GastrExtub
Status: Terminated | Type: Observational
Why Stopped: Patient enrollment difficulties
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1249; 2021-A03130-41 (Other: ID-RCB)
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Fasting; Pediatric ALL; Aspiration
Keywords: Fasting; Extubation; Pediatric critical care; Gastric ultrasound; Aspiration
MeSH Terms: conditions — Fasting; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill children ready for extubation: Children admitted to a paediatric intensive care unit, invasively ventilated and intubated, enterally fed and presenting with a clinical condition allowing for extubation. 45 children will be included.
  Interventions: Other: Gastric ultrasound

INTERVENTIONS:
Other: Gastric ultrasound — Assessment of gastric content with gastric ultrasound monitoring: gastric ultrasounds will be performed in eligible children, when enteral feeding is stopped for planned extubation, and repeated 6 hours after, at extubation and every hour between feeding interruption and extubation. The stomach will be classified as empty or full according to PERLAS criteria. In total, 8 gastric ultrasounds will be performed over a period of 12 hours.

SUMMARY:
Nearly half of critically ill children are intubated and enterally fed according to recent guidelines. However, no evidence-based recommendation are available regarding fasting times prior to extubation.

When an extubation is planned, children do not always present with normal neurological status yet, and are at risk of vomiting and aspiration. Extubation may also fail and require re-intubation with similar risks. Thus, pre-operative fasting guidelines are often transposed to the paediatric critical care setting, aiming for an empty stomach at extubation, with perceived decreased risks of aspiration. However, the gastric and gut motility pathophysiology is significantly different in critically ill children (frequent gastroparesis, liquid continuous feeding, etc.) compared to planned surgery children. The extrapolation of practice validated in the latter population may be inadequate. The stomach may be empty more or less rapidly than expected, leading to unnecessary prolonged fasting times or inappropriately short fasting times respectively.

Gastric ultrasounding monitoring may help assessing gastric content prior to extubation.

Investigators hypothesise gastric content clearance may be different in critically ill children prior to extubation, compared to pre-operative paediatric guidelines for elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 17 year old children admitted to pediatric intensive care unit
* intubated (oral or nasal tracheal tube)
* gastric enteral feeding affording at least 25% of the nutritional target (estimated with Schofield equations)
* No opposition from one of the 2 parents (or legal representatives)

Exclusion Criteria:

* anatomical anomaly of the stomach location (e.g. post surgery)
* Difficult access to perform gastric ultra-sounding (drains, plasters, dressings etc.)
* mobilization to right lateral decubitus at risk

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 45 critically ill children (meeting inclusion criteria and respecting exclusion criteria), will be recruited in a single pediatric intensive care unit, if they are intubated and enterally fed on a gastric tube.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Percentage of critically ill children presenting with a full stomach 6 hours after enteral feeding interruption for planned extubation | 12 hours following the inclusion
  Percentage of critically ill children presenting with a full stomach (according to PERLAS criteria) 6 hours after enteral feeding interruption for planned extubation. Gastric emptiness is assessed with gastric ultrasounding, depicting gastric content (empty versus full). Antral diameter will also be measured and gastric volume will be calculated to allow classifying gastric content according to PERLAS criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Paediatric intensive care Unit - Hopital Femme Mère Enfant - Hospices Civils de Lyon, Bron, France